CLINICAL TRIAL: NCT03356548
Title: Study of the Association Between Transferrin Saturation and Asthenia in Hemochromatosis
Brief Title: Transferrin Saturation and Asthenia in Hemochromatosis
Acronym: HEMOSAT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3067_HEMOSAT
Record Dates: First submitted 2017-11-16; First posted 2017-11-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hemochromatoses, Genetic
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study.

DETAILED DESCRIPTION:
The linked HFE genetic hemochromatosis (C282Y mutation in the homozygous state) is the most common form of genetic iron overload.

Its treatment is based on bloodletting, and takes place in 2 phases, according to the recommendations of the High Authority of Health (HAS). The first phase, called induction, aims to achieve ferritinemia <50 by performing weekly bleeds.

The second phase, called maintenance, aims to maintain this ferritinemia <50 by performing bleeding every 1 to 6 months depending on the case.

The treatment is therefore according to the current recommendations only adapted according to ferritinemia, and not according to the effectiveness on the functional symptoms. However, some patients report persistent asthenia during maintenance treatment, despite ferritin levels <50. This could reflect an incomplete control of their disease, and leads us to raise two points:

* It is known that in some subjects, the Transferrin Saturation Coefficient remains high, despite ferritinemia <50; it is also known that this elevation of the Transferrin Saturation Coefficient may be accompanied by a rise in circulating free iron, which is toxic for the organism1.
* The asthenia observed in some patients in the maintenance phase could be linked to a high rate of Transferrin Saturation Coefficient.

Our objective is to evaluate, in patients homozygous C282Y in maintenance phase, the association between quality of life and Transferrin Saturation Coefficient .

ELIGIBILITY:
* Inclusion criteria:

  * homozygous C282Y ;
  * in the maintenance phase for at least 6 months ;
  * follow-up at Rennes University Hospital ;
  * patient who has not expressed his opposition to participate in the study.
* Exclusion criteria:

  * Permanent: any cause of modification of the CST unrelated to hemochromatosis (chronic inflammatory disease, excessive consumption of alcohol ...) ;
  * Temporary: infectious syndrome within 7 days before bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with genetic hemochromatosis HFE
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire SF 36 | Through study completion, an average of 3 months
Biological markers : Transferrin Saturation Coefficient | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice LAINE, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Britain, France